CLINICAL TRIAL: NCT02750644
Title: Post Approval Non-randomized Double-arm Prospective Open Label Follow-up Trial on Carotid Stenting Using MOMA Proximal Embolic Cerebral Protection Device in Patients With High Risk vs Standard Risk for Open Carotid Endarterectomy(REALTrial)
Brief Title: Postapproval Trial On Carotid Stenting in Patients With High Risk Vs Standard Risk for Open Carotid Endarterectomy(REAL)
Acronym: REAL
Status: Completed | Type: Observational
Sponsor: Joaquin de Haro, M.D. (Other)
Responsible Party: Sponsor-Investigator, Joaquin de Haro, M.D., Joaquin de Haro, M.D., Vascular Research Unit Principal Investigator, Hospital Universitario Getafe
Organization: Hospital Universitario Getafe (Other)
Other Study IDs: REAL
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High-risk: Patients with atherosclerotic carotid disease with (1) severe comorbidity (class III/IV congestive heart failure, class III/IV angina, coronary disease involving ≥ 2 major vessels, left ventricular ejection fraction ≤ 30%, myocardial infarction, severe pulmonary disease, severe renal failure) and (2) Technical/challenging anatomical criteria (previous neck surgery, cervical irradiation, contralateral carotid occlusion, post-endarterectomy restenosis, inaccessible lesions or tracheotomy).
- Standard-risk: Patients with atherosclerotic carotid disease without (1) severe comorbidity (class III/IV congestive heart failure, class III/IV angina, coronary disease involving ≥ 2 major vessels, left ventricular ejection fraction ≤ 30%, myocardial infarction, severe pulmonary disease, severe renal failure) and (2) Technical/challenging anatomical criteria (previous neck surgery, cervical irradiation, contralateral carotid occlusion, post-endarterectomy restenosis, inaccessible lesions or tracheotomy).

SUMMARY:
Until the irruption of the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST), carotid stenting (CAS) has been mainly offered to those patients considered at "high risk" for open carotid endarterectomy (CEA) based on the available data from large randomized clinical trials. "High risk" has been defined as (1) patients with severe comorbidity (class III/IV congestive heart failure, class III/IV angina, coronary disease involving ≥ 2 major vessels, left ventricular ejection fraction ≤ 30%, myocardial infarction, severe pulmonary disease, severe renal failure) and (2) Technical/challenging anatomical criteria (previous neck surgery, cervical irradiation, contralateral carotid occlusion, post-endarterectomy restenosis, inaccessible lesions or tracheotomy). Several recent studies have called medical "high-risk" into question for CAS indication.

The purpose of this study is to evaluate the safety and perioperative and long-term effectiveness in patients with significant carotid artery stenosis with "high-risk" criteria (for CEA) treated with carotid stenting and proximal protection device (MOMA®) compared to patients with standard-surgical-risk features.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients who have a transient ischemic attack, amaurosis fugax, or minor nondisabling stroke in the distribution of the study artery within 180 days of inclusion and have been shown carotid artery stenosis ≥50% by angiography, ≥70% by ultrasound, or ≥70% by CT angiography or MR angiography if ultrasound is 50% to 69%
* Asymptomatic patients who have carotid artery stenosis of ≥60% by angiography, ≥70% by ultrasound, or ≥80% by CT angiography or MR angiography if ultrasound is 50% to 69%

Exclusion Criteria:

* Patient is unable to respond to external questions and stimuli and to exert a pressure with the contralateral hand
* Patient has an myocardial infarction within 72 hours prior to carotid stenting
* Patient has a major residual neurological deficit (stroke scales: Barthel ≤ 60, NIH ≥ 15 or Rankin >3) at pre-procedure neurological exam
* Patient had a transient ischemic attack (TIA) or amaurosis fugax within 48 hours prior to index procedure
* Patient had a stroke or retinal artery occlusion within 1 month prior to index procedure
* Patient has severe chronic renal failure (creatinine > 2.5mg/dL)
* The target carotid artery is completely occluded
* The common carotid artery ostium has stenosis that required treatment
* The presence of ipsilateral intracranial stenosis that requires treatment
* The inability to position a stiff 0.035" guidewire in the external carotid artery
* Contralateral occlusion of internal carotid artery and vertebral arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Internal carotid stenosis symptomatic patients who have a transient ischemic attack, amaurosis fugax, or minor nondisabling stroke in the distribution of the study artery within 180 days of inclusion and have been shown carotid artery stenosis ≥50% by angiography, ≥70% by ultrasound, or ≥70% by CT angiography or magnetic resonance (MR) angiography if ultrasound is 50% to 69%. Asymptomatic patients who have carotid artery stenosis of ≥60% by angiography, ≥70% by ultrasound, or ≥80% by CT angiography or MR angiography if ultrasound is 50% to 69%.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2005-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
all major adverse events | through 30-day follow-up or thereafter up to 4 years
  the composite rate of all major adverse events (MAE), including death, stroke, and Myocardial Infarction, through 30-day follow-up or thereafter up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin De Haro, MD, Principal Investigator — Hospital Universitario Getafe

IPD SHARING:
Plan to Share IPD: Undecided